CLINICAL TRIAL: NCT04331379
Title: Effectiveness of Nasal-alar Elevator (NE) Combined With Taping Vs. Taping Alone on Improving the Nose Esthetics and Maxillary Arch Dimensions in Infants With Unilateral Complete Cleft Lip and Palate: A Randomized Clinical Trial
Brief Title: Effectiveness of Nasal-alar Elevator Combined With Taping Vs. Taping Alone on Improving the Nose Esthetics and Maxillary Arch Dimensions in Infants With Unilateral Complete Cleft Lip and Palate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Abd El-Ghafour, Lecturer of Orthodontics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Cleft Lip and Palate
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal Elevator (Experimental)
  Interventions: Device: Nasal Elevator
- Taping Alone (Active Comparator)
  Interventions: Device: Taping Alone

INTERVENTIONS:
Device: Nasal Elevator — A device aiming to elevate the clefted nostril extraorally and fixed on the forehead.
  Arms: Nasal Elevator
Device: Taping Alone — Horizontal tape alone.
  Arms: Taping Alone

SUMMARY:
This randomized trial is designed to assess the effectiveness of nasal elevator as a presurgical infant orthopedics on improvement of nose esthetics vs taping alone.

ELIGIBILITY:
Inclusion Criteria:

* Infants with age range from 1-30 days.
* Unilateral complete cleft lip and alveolus.
* Medically free subjects.
* Both males and females.
* Cleft gap more than 10 mm.

Exclusion Criteria:

* Patients older than 30 days.
* Syndromic patients with other defects in addition to cleft lip and palate.
* Patients with bilateral cleft lip and palate.
* Incomplete Cleft lip.
* Patient with previous surgical lip repair or adhesion.
* Patients with previous presurgical infant orthopedic treatment.
* Medically compromised patients.
* Cleft gap distance less than 10mm

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Nasal Esthetics | 3 months
  Nasal esthetics will be following Dr Farkas' measurements and it will be carried out as linear and angular measurements on standardized photographs. it will be measured using photoshop software.
Maxillary arch changes | 3 months
  Different maxillary arch dimensions (e.g. cleft and arch widths and symmetry) will be measured virtually on digital models in mm using 3shape software.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided